CLINICAL TRIAL: NCT01802541
Title: Effect of Diacylglycerol Oil on Risk Factors of Type 2 Diabetes and Complicating Disease, and Mechanism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Duo li, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: P031217
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Insulin Sensitivity; Type 2 Diabetes; Cardiovascular Disease
Keywords: diacylglycerol oil; insulin sensitivity; type 2 diabetes; cardiovascular disease; risk factors
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Diglycerides; Triglycerides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAG oil (Experimental)
  Interventions: Dietary Supplement: diacylglycerol oil
- TAG oil (Placebo Comparator)
  Interventions: Dietary Supplement: triacylglycerol oil

INTERVENTIONS:
Dietary Supplement: diacylglycerol oil
  Arms: DAG oil
Dietary Supplement: triacylglycerol oil
  Arms: TAG oil

SUMMARY:
Diacylglycerol oil has been shown to lower postprandial and fasting serum triacylglycerol levels and reduce body fat. The investigators hypothesize that replacing dietary fat with diacylglycerol oil reduces excess body fat in type 2 diabetic patients and that diacylglycerol oil has a beneficial effect on cardiovascular risk factors in Chinese type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic patients, blood sugar levels were stabilized between 7.0-10.0 mmol/L
2. Male, aged 40 - 70 years old, Female, aged post-menopausal - 70 years old.
3. Overweight/obese patients (BMI 25 - 40 kg/m2)
4. Currently under diet therapy for diabetes mellitus
5. Understands the procedures and willing to participate in the study

Exclusion Criteria:

1. Patients who unwilling to give informed consent
2. Type 1 diabetic patients
3. Familial hyperlipemia patients or blood triacylglycerol concentration > 400 mg/dl
4. Patients with a history of cardiovascular disease and/or arteriosclerotic disease
5. Patients with a history of cerebrovascular disease
6. Patients with serious hepatic disease and/or renal disease
7. Patients with malignancy
8. Participation in another clinical study within 30 days prior to screening period.
9. Has a condition the doctor in charge believes would interfere with evaluation of the subject, or may put subject at undue risk

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
insulin resistance | 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Duo Li, Ph.D., Principal Investigator